CLINICAL TRIAL: NCT02190630
Title: A Prospective Randomised Controlled Trial Investigating the Skeletal and Dental Effects of a Removable Brace That Works on the Upper and Lower Teeth at the Same Time Worn Part Time Versus Full Time
Brief Title: Study to Measure the Effect of Part Time Versus Full Time Orthodontic Appliance Wear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Mary University of London (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ReDA Ref: 009038
Record Dates: First submitted 2014-03-12; First posted 2014-07-15 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-09

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part time (12hour) wear (Active Comparator): the' Modified Clark Twin Block' will be worn part time
  Interventions: Device: Modified Clark Twin Block
- Full time (24hour) wear (Active Comparator): the ' Modified Clark Twin Block' will be worn full time
  Interventions: Device: Modified Clark Twin Block

INTERVENTIONS:
Device: Modified Clark Twin Block — The Modified Clark Twin Block is a type of functional orthodontic appliance used to posture the lower jaw forward to treat discrepancies between the upper and lower jaw bones
  Other Names: Clark Twin Block; Twin Block; Functional Appliance

SUMMARY:
The aim of this study is to assess skeletal (bone) and dental (teeth) changes occurring following wear of a twin block functional appliance (removable brace which postures the lower jaw forward to improve a discrepancy between the upper and lower jaw) for differing time periods.

DETAILED DESCRIPTION:
Functional appliances are ordinarily worn full time in adolescence between 11 and 14 years with a discrepancy between their upper and lower jaws. The reason it is worn between these ages is to avail of the pre pubertal growth spurt, evidence for full time wear is merely empirical.If this appliance only had to be worn part time it would have a significant change in orthodontics in terms of patient acceptance and compliance.The investigators plan on recruiting 84 patients to the study and these subjects will be referred from hospital colleagues. The investigators will randomly allocate the subjects into 2 groups, Group 1 will wear the appliance Full Time(24hours), group 2 will wear the appliance part time(12hours).

The study will be conducted in the Dental Institute at the Royal London Hospital, this hospital setting will be the sole site.

The study will last for 15 months from the time the last patient is recruited. Participants will undergo an initial records appointment where a radiograph and clinical measurements will be taken followed by 12 months of functional appliance treatment where the patient will be reviewed at 6-8weekly intervals and clinical measurements taken.A final radiograph will be taken at 15months.

ELIGIBILITY:
Inclusion Criteria:

* Class II div 1 malocclusion(upper front teeth lying more forward than lower front teeth with upper front teeth proclined),
* Overjet(horizontal difference between upper and lower front teeth) measuring minimum of 7mm,
* Male subjects 12--14 years at the start of treatment,
* Female subjects 11--13 years at start of treatment,
* Willingness of the patient and parent to participate in the study.

Exclusion Criteria:

* No previous orthodontic treatment
* No relevant medical history or craniofacial syndrome

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2013-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
remaining overjet measured with an orthodontic ruler | outcome measure will be assessed after 12 months appliance wear and after a 3 month relapse period
  the initial overjet will compared to the final overjet following 12 months of appliance treatment, and 3 months of relapse. overjet will be measured with an orthodontic ruler at every review appointment
Cephalometric Changes | Outcome will be assessed after 12m of appliance wear and after 3 months of settling.
  Both linear and angular cephalometric changes will be assessed over this timeframe.

SECONDARY OUTCOMES:
Comparison of subjective and objective measures of appliance wear | 12 months of appliance wear
  Subjective (patient completed time charts) and objective (theramon micro-sensor) measures of wear will be assessed over 12months of appliance wear.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Counihan, BDS, Principal Investigator — Queen Mary University of London; Jeet Parekh, BDS, Principal Investigator — Queen Mary University of London
Locations (1):
- Dental Insitiute Royal London Hospital, London, London, United Kingdom

REFERENCES:
- [Derived] Parekh J, Counihan K, Fleming PS, Pandis N, Sharma PK. Effectiveness of part-time vs full-time wear protocols of Twin-block appliance on dental and skeletal changes: A randomized controlled trial. Am J Orthod Dentofacial Orthop. 2019 Feb;155(2):165-172. doi: 10.1016/j.ajodo.2018.07.016. PMID 30712687